CLINICAL TRIAL: NCT02130999
Title: A Single Dose, Open-Label, Randomized Two-Period Crossover Study in Healthy Young Subjects to Assess the Absolute Bioavailability of Tasimelteon (HETLIOZ™)
Brief Title: Open Label Study to Assess the Absolute Bioavailability of Tasimelteon (HETLIOZ™)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VP-VEC-162-4101
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Non-24-Hour-Sleep-Wake Disorder
Keywords: Non-24; absolute bioavailability; tasimelteon; Hetlioz™
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — tasimelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental): * Single oral dose of tasimelteon 20 mg on Day 1
  * Single I.V. dose of tasimelteon 2 mg on Day 6
  Interventions: Drug: tasimelteon 20 mg capsule; Drug: tasimelteon 2 mg I.V.
- Sequence B (Experimental): * Single I.V. dose of tasimelteon 2 mg on Day 1
  * Single oral dose of tasimelteon 20 mg on Day 6
  Interventions: Drug: tasimelteon 20 mg capsule; Drug: tasimelteon 2 mg I.V.

INTERVENTIONS:
Drug: tasimelteon 20 mg capsule
  Other Names: Hetlioz™ 20 mg
Drug: tasimelteon 2 mg I.V.

SUMMARY:
Hetlioz™ (tasimelteon) is used in the treatment of Non-24-Hour-Sleep-Wake Disorder (Non-24). Non-24 is very common in people who are totally blind because light can not reset their body clock. This causes the internal sleep-wake cycle to be out of sync with the 24-hour day-night. Non-24 is a serious, chronic circadian rhythm disorder in the blind that causes nighttime sleep problems and a wide range of daytime difficulties, including an overwhelming urge to nap.

Tasimelteon will be given in two ways; orally (by mouth) as a 20 mg capsule and intravenously (I.V.) by infusion through a catheter (not an injection) into a vein. The oral administration is approved by the FDA. The I.V. administration is considered investigational as it has not been approved by the FDA. This will be the first time tasimelteon will be given to humans by intravenous (I.V.) injection.

The purposes of this research study are to:

* assess how quickly a single 20 mg oral dose of tasimelteon is absorbed into the body;
* evaluate the single-dose pharmacokinetics of tasimelteon after a single 20 mg oral dose and after a single 2 mg I.V. dose;
* evaluate the single-dose pharmacokinetics of tasimelteon metabolites after a single 20 mg oral dose and after a single 2 mg I.V. dose;
* evaluate the safety and tolerability of a single 20 mg oral dose of tasimelteon; and
* evaluate the safety and tolerability of a single 2 mg I.V. dose of tasimelteon.

Pharmacokinetics (PK) is the study of how a drug is absorbed, distributed, metabolized, and eventually eliminated by the body. Pharmacokinetics is what the body does to the drug. Blood samples will be taken throughout the study for PK analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18 - 55 years, inclusive;
2. Non-smokers [abstinence from smoking for at least 6 months before the screening visit] and test negative for cotinine at screening and baseline;
3. Subjects with Body Mass Index (BMI) of ≥18 and ≤25 kg/m2 (BMI = weight (kg)/ [height (m)]2);
4. Males, non-fecund females (i.e., surgically sterilized, if procedure was done 6 months before screening or subject is postmenopausal, without menses for 6 months before screening), or females of child-bearing potential using an acceptable method of birth control for a period of 35 days before the first dosing, and females must have a negative pregnancy test at the screening and baseline visits; Note 1: Acceptable methods of birth control include any one of the following: abstinence, vasectomized sexual partner, hormonal methods (i.e. pill, hormonal IUD, Depo-Provera, implants, patch, intravaginal device [NuvaRing]), intrauterine device (IUD [copper banded coils]), diaphragm, cervical cap, or condom with spermicidal jelly or foam
5. Vital signs (after 3 minutes resting in a semi-supine position) which are within the ranges shown below:

   1. Body temperature between 35.0-37.5 °C;
   2. Systolic blood pressure between 90-150 mmHg;
   3. Diastolic blood pressure between 50-95 mmHg;
   4. Pulse rate between 50-100 bpm.
6. Ability and acceptance to provide written informed consent;
7. Willing and able to comply with study requirements and restrictions;
8. Subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, clinical laboratory tests and urinalysis;

Exclusion Criteria:

1. History of recent (within six months) drug or alcohol abuse as defined in DSM-V, Diagnostic Criteria for Drug and Alcohol Abuse or evidence of such abuse as indicated by the laboratory assays conducted during the Screening Visit or at Baseline;
2. Any major surgery within three months of the first Baseline visit or any minor surgery within one month;
3. History or current evidence of cardiovascular, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction or psychiatric disease judged by the Investigator to be clinically significant;
4. Subjects who are currently considered a suicide risk, any subject who has ever made a suicide attempt, or those who are currently demonstrating active (within the past 6 months) suicidal ideation as deemed by the Columbia Suicide Severity Rating Scale (C-SSRS);
5. Any condition requiring the regular use of medication except those listed in Section 8.2;
6. Exposure to any investigational drug, including placebo, within 30 days or 5 half-lives (whichever is longer) of baseline
7. Exposure (within 2 weeks of Day -1) to any over-the-counter medications including melatonin, dietary supplements and/or herbal remedies, except those listed on Section 8.2;
8. Treatment with any drug known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) during the 60 days preceding the Screening visit;
9. History of intolerance and/or hypersensitivity to tasimelteon, and/or drugs similar to tasimelteon including melatonin;
10. Donation or loss of 400 mL or more of blood within one month prior to the Baseline Visit;
11. Significant illness within the two weeks prior to Baseline;
12. Pregnant or lactating females;
13. History of porphyria or liver disease and/or positive for one or more of the following serological results:

    1. A positive hepatitis C antibody test (anti-HCV)
    2. A positive hepatitis B surface antigen (HBsAg)
    3. A positive HIV test result
14. Use of any food or beverage containing grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g. kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard greens) and charbroiled meats for at least 2 weeks before the Baseline Visit until the end of the study;
15. Inability to be venipunctured and/or tolerate venous access;
16. Previous participation in a BMS-214778, VEC-162, or tasimelteon study;
17. Subjects who are unable to read or speak English;
18. Any other sound medical reason as determined by the clinical Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A: * Single oral dose of tasimelteon 20 mg on Day 1
  * Single I.V. dose of tasimelteon 2 mg on Day 6
  tasimelteon 20 mg capsule
  tasimelteon 2 mg I.V.
- Sequence B: * Single I.V. dose of tasimelteon 2 mg on Day 1
  * Single oral dose of tasimelteon 20 mg on Day 6
  tasimelteon 20 mg capsule
  tasimelteon 2 mg I.V.
Period: Overall Study
Arm/Group | Sequence A | Sequence B
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Number of Baseline Participants: 14 subjects total participated in the study
Arm/Group | Overall Number of Baseline Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Body Mass Index [Mean (Standard Deviation); unit: (kg/m^2)] | 22.8 (1.8)
Weight [Mean (Standard Deviation); unit: (kg)] | 63.6 (8)
Height [Mean (Standard Deviation); unit: (cm)] | 166.6 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Bioavailability After a Single Oral Dose of Hetlioz™(Tasimelteon) 20mg
Description: The absolute bioavailability (F) of tasimelteon will be estimated from the dose-corrected AUC(inf) after oral and I.V. administration using an analysis of variance (ANOVA) model with treatment, period, sequence, and subject within sequence as the classification variables, using natural log-transformed data. The geometric mean ratio (GMR), oral-to-I.V., and its associated 90% confidence interval (CI) will be used as the estimate of F and its variability.
Time Frame: pre-dose, -0.125, 0, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Measure: Geometric Mean (90% Confidence Interval); unit: Geometric Mean Ratio (%)
Arm/Group | Absolute Bioavailability
Number analyzed (Participants) | 14
Geometric Mean Ratio (%) | 38.3 [26.9 to 54.3]

2. Secondary Outcome: Cmax of Tasimelteon After a Single 20 mg Oral Dose and After a Single 2 mg I.V. Administration.
Description: Cmax of tasimelteon will be compared when given orally or administered as an I.V.
Time Frame: pre-dose, -0.125, 0, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oral (20 mg) | IV (2 mg)
Number analyzed (Participants) | 14 | 14
ng/mL | 260 (189) | 82.2 (20.5)

3. Secondary Outcome: AUC (Inf) of Tasimelteon After a Single 20 mg Oral Dose and After a Single 2 mg I.V. Administration.
Description: AUC (inf) of Tasimelteon will be compared when given orally or administered as an I.V.
Time Frame: pre-dose, -0.125, 0, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Measure: Mean (Standard Deviation); unit: (h*ng/mL)
Arm/Group | Oral (20 mg) | IV (2 mg)
Number analyzed (Participants) | 14 | 14
(h*ng/mL) | 358 (271) | 71.6 (23.9)

4. Secondary Outcome: T1/2 of Tasimelteon After a Single 20 mg Oral Dose and After a Single 2 mg I.V. Administration.
Description: T1/2 of tasimelteon will be compared when given orally or administered as an I.V.
Time Frame: pre-dose, -0.125, 0, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours pos-dose
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Oral (20 mg) | IV (2 mg)
Number analyzed (Participants) | 14 | 14
hour | 1.06 (0.23) | 1.02 (0.23)

5. Secondary Outcome: Total Clearance of Tasimelteon After a Single 20 mg Oral Dose and After a Single 2 mg I.V. Administration.
Description: CL of tasimelteon will be compared when given orally or administered as an I.V.
Time Frame: pre-dose, -0.125, 0, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Measure: Mean (Standard Deviation); unit: (mL/min)
Arm/Group | Oral (20 mg) | IV (2 mg)
Number analyzed (Participants) | 14 | 14
(mL/min) | 2241 (3592) | 505 (135)

6. Secondary Outcome: Cmax of Tasimelteon's Metabolites After an Oral and I.V. Dose of Tasimelteon
Description: The mean +/- SD for the Cmax of tasimelteon's metabolites after a single 20 mg oral dose of tasimelteon and after a single 2 mg I.V. administration of tasimelteon
Time Frame: pre-dose, -0.125, 0, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oral (20 mg) | IV (2 mg)
Number analyzed (Participants) | 14 | 14
ng/mL
  M9 | 303 (94.3) | 16.4 (6.16)
  M11 | 53.2 (16.14) | 3.7 (1.25)
  M12 | 113 (30.8) | 7.31 (2.49)
  M13 | 370 (105) | 29 (11.7)

7. Secondary Outcome: AUC(Inf) of Tasimelteon's Metabolites After a Single Oral and I.V. Dose
Description: The mean +/- SD for the AUC(inf) of tasimelteon's metabolites after a single 20 mg oral dose of tasimelteon and after a single 2 mg I.V. administration of tasimelteon
Time Frame: pre-dose, -0.125, 0, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: Only 11 subjects could be analyzed for M11.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Oral (20 mg) | IV (2 mg)
Number analyzed (Participants) | 14 | 14
h*ng/mL
  M9 | 400 (139) | 30.3 (10.3)
  M11 | 125 (43.7) | 12.2 (4.40)
  M12 | 619 (364) | 43.8 (25.4)
  M13 | 431 (152) | 38.2 (13)

8. Secondary Outcome: Metabolite-to-parent AUC(Inf) Ratios After Oral Administration of a Single 20 mg Dose and IV Administration of a Single 2 mg Dose of Tasimelteon
Description: Comparison of the metabolite-to-parent AUC(inf) ratios for the oral and IV routes.
Time Frame: pre-dose, -0.125, 0, 0.083, 0.167, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Measure: Mean (Standard Deviation); unit: metabolite to parent AUC (inf) ratios
Arm/Group | Oral (20 mg) | IV (2 mg)
Number analyzed (Participants) | 14 | 14
metabolite to parent AUC (inf) ratios
  M9 | 1.98 (2.65) | 0.39 (0.12)
  M11 | 0.51 (0.35) | 0.16 (0.03)
  M12 | 2.04 (0.93) | 0.54 (0.15)
  M13 | 1.72 (1.12) | 0.51 (0.14)

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse event per treatment arm and overall.
Time Frame: From Baseline to End of Study; Day 5 (± 2 days).
Measure: Number; unit: participants
Arm/Group | Tasimelteon 20mg Oral | Tasimelteon 2mg IV | All Subjects
Number analyzed (Participants) | 14 | 14 | 14
participants
  vomiting | 0 | 1 | 1
  headache | 1 | 1 | 2
  Somnolance | 1 | 0 | 1

10. Other Pre Specified Outcome: Number of Participants That Reported Suicidal Ideation, Suicidal Behavior, or Suicide Attempts.
Description: Number of Participants that reported suicidal ideation, suicidal behavior, or suicide attempts per treatment arm and overall.
Time Frame: Baseline to End of Study Day 5 (± 2 days).
Measure: Number; unit: participants
Arm/Group | Tasimelteon 20mg Oral | Tasimelteon 2mg IV | All Subjects
Number analyzed (Participants) | 14 | 14 | 14
participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Tasimelteon 20mg Oral | Tasimelteon 2mg IV | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/14 | 1/14 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tasimelteon 20mg Oral (N=14) | Tasimelteon 2mg IV (N=14) | All Subjects (N=14)
headache (Nervous system disorders) | 1 | 1 | 2
sommolence (Nervous system disorders) | 1 | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days